CLINICAL TRIAL: NCT02360826
Title: Pharmacokinetics of Pravastatin and Simvastatin in Pediatric Dyslipidemia Patients: Clinical Impact of Genetic Variation in Statin Disposition
Brief Title: Statin Distribution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Jon Wagner, DO, Children's Mercy Hospital Kansas City
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13CRP1711002
Record Dates: First submitted 2013-09-03; First posted 2015-02-11 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Drug Distribution
MeSH Terms: interventions — Pravastatin; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pravastatin (Experimental): Pravastatin 20mg tablet (age 8-13 years), 40mg tablet (>14 years); 1 time dose given per oral at at the start of the study day.
  Interventions: Drug: Pravastatin
- Simvastatin (Experimental): Simvastatin 10mg tablet (ages 8-13 years), 20mg tablet (>14 years); 1 time dose given per oral at the start of the study day.
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Pravastatin
  Arms: Pravastatin
Drug: Simvastatin
  Arms: Simvastatin

SUMMARY:
Anticipating an increased use of statins in children and adolescents, it is imperative that we understand the genetic and developmental characteristics affecting the pharmacokinetics and pharmacodynamics of statins in childhood and adolescence. Simply extrapolating pediatric dosing guidelines from adult dose-exposure-response relationships fails to recognize the potential impact of growth and development in pediatric patients, which may have important clinical implications for drug efficacy or toxicity. Current evidence indicates that genetic variation in the SLCO1B1 transporter is important for statin disposition and toxicity in adults. The ontogeny of SLCO1B1 during human growth and development has not been well characterized, and limited pediatric data indicate that the genotype-phenotype relationship in children is the opposite of that observed in adults. Therefore, investigating the relative roles of SLCO1B1 ontogeny and genetic variation in statin disposition and response is key to determining the age at which the statin dose-exposure-response relationship mimics adults, and has important implications for other medications transported by the SLCO1B1 protein.

As the first step in this process, our specific aims for the current investigation are 1) to determine the effect of genetic variation of SLCO1B1 on the pharmacokinetics of pravastatin and simvastatin by comparing Cmax, AUC and elimination between children and adolescents with 2 functional SLCO1B1 alleles and those with one or more variant alleles, and 2) to determine if the magnitude of the genetic effect on pravastatin pharmacokinetics (defined as Cmax, AUC and elimination) is equivalent to the effect on simvastatin pharmacokinetics. As a secondary aim, Cmax and AUC of pravastatin and simvastatin will be compared between children and adolescents for each genotype group. These results will be utilized to determine the sample size necessary to adequately power future studies characterizing the role of ontogeny on statin disposition.

The ultimate goal of this proposed investigation is to establish the role of genetic variation in key transporters on the dose-exposure relationship of two commonly used statin drugs in children. This study is the first step in a series of investigations aimed at determining the mechanisms behind variations in physiologic response, clinical efficacy and significant adverse effect risk that surround the statin drugs in children and adolescents.

DETAILED DESCRIPTION:
The ultimate goal of this proposed investigation is to establish the role of genetic variation and development in key transporters on the dose-exposure relationship of two commonly used statin drugs in children. This study is the first step in a series of investigations aimed at determining the mechanisms behind variations in physiologic response, clinical efficacy and significant adverse effect risk that surround the statin drugs in children and adolescents.

Research Design and Methods

1. Trial Design 1.1. Investigational Agents Pravastatin 20 mg tablet (ages 8-13 years), 40 mg tablet (>14 years) Simvastatin 10 mg tablet (ages 8-17), 20mg (>17 years) Commercial supplies of pravastatin and simvastatin that are FDA approved for use in pediatric dyslipidemia will be used. Pravastatin and simvastatin from the same source and lot will be used for all subjects. The doses designated above are chosen according to previous adult and pediatric data 26, 28-32, 41 and are consistent with current labeling for pravastatin and simvastatin. Although fixed doses within a pre-specified age range will be used, dose data will be analyzed corrected for weight (mg/kg) based on the patient's weight at time of dosing.

1.2. Risk/Benefits All subjects with a LDL >130mg/dl (95% percentile) will be eligible for this study, consistent with current clinical criteria for statin therapy. The risks associated with participation in this single-dose pharmacokinetic study are expected to be minimal given the known adverse event profile for the study articles and also, the limited exposure. The most common mild adverse effects of statins are headache, myalgia, and gastrointestinal symptoms (abdominal pain, dyspepsia, diarrhea, constipation). However, in children these adverse effects occur with the same frequency as placebo 14, 15, 18. Rare adverse effects include elevation of hepatic transaminases and myopathy, but these are generally observed with chronic treatment. Furthermore, no cases of hepatic failure with statins have been reported to date 52. There is also a small risk associated with placement of the intravenous (IV) catheter that will be used to draw serial blood samples for pharmacokinetic analysis and screening/safety labs. Finally, there is the risk of loss of confidentiality for the participating subjects. Methods to protect PHI and data handling are specifically outlined in the CMH CPR protocol Sections 4 & 5 (CMH IRB# 12040220). All of the above risks associated with this non-therapeutic clinical trial are minimal.

There is no direct benefit to participating subjects, although there may be benefit for children in the future as it is expected that the information to be gained from the study can be generalized to the larger population of pediatric patients who may require statin treatment. The purpose of the study is to determine how genetic variation impacts pravastatin and simvastatin plasma concentrations following recommended doses of the drug in a patient population that has not previously been studied. Thus, with this knowledge, future protocols could subsequently be developed to effectively "personalize" dosing for pediatric subjects with the aforementioned SNPs who are taking pravastatin or simvastatin, thereby improving efficacy and safety for the individual patient.

1.3. Study Design/Type This will be a single center, open label, randomized, cross-over study in patients with dyslipidemia comparing the pharmacokinetics of pravastatin and simvastatin, in patients with greater than or equal to one variant allele in the SLCO1B1 gene (-11187 and/or c.521) to patients with the wild-type/wild-type genotype.

1.4. Population Sample The CMH Cardiology Pharmacogenomics Repository (CPR) (CMH IRB# 12040220) database will be accessed to determine subjects meeting inclusion criteria. Once the target population and an equal set of age-, sex- and Tanner Stage-matched controls are identified, the patients will be invited to participate in a single center, open label, randomized, cross-over, pharmacokinetic study of pravastatin and simvastatin.

1.5. Subject Recruitment Once a target population and an equal set of age- and sex-matched controls are identified from the CPR, prospective participants will be informed about the study. Initial contact will occur by way of a prepared telephone script. Those that agree to participate will be scheduled for a visit to the CMH Clinical Research Unit for a screening visit. At this visit, the study will be explained to the patient/patient's family, permission/assent/consent will be obtained, a physical examination (including Tanner staging), and screening laboratory testing will be performed. Participants for whom permission/assent/consent has been obtained and inclusion criteria are met, will be scheduled to come back to the CMH Clinical Research Unit within 6 to 14 days for the first study drug day.

1.6. Subject Withdrawal Participation in the pharmacokinetic trial of pravastatin and simvastatin is completely voluntary. As part of the informed permission/assent/consent process; subjects are informed that they can withdraw their permission/assent/consent at any time. If at any time, study subjects have social, philosophical, religious or family concerns related to the study, they may decide to withdraw permission/assent/consent.

A study subject or an authorized third party (PCP) may revoke permission/assent/consent at anytime. The request to revoke permission/assent/consent may be made verbally or in writing and addressed to study personnel (as indicated in the permission/assent/consent form). Study personnel will take appropriate steps to respect the will of the study subject and ensure that the study subject is able to withdraw without having a compromise in personal integrity or medical evaluation/treatment. In the event permission/assent/consent to continue is withdrawn after partial collection of samples or data, only existing data will be analyzed and tabulated. The subject can be withdrawn from the study by the investigators, if at any point, in the judgment of the investigators, that the subject's continued participation may be associated with the production of unanticipated risks (e.g., a late onset hypersensitivity reaction following administration of the study article).

1.7. Subject Study Visits The study will involve three total visits. One screening visit and 2 drug study day visits.

Screening Visit (Approximately 1 hour) -Upon arrival for the screening visit, the study will be reviewed in depth with the participating subject and subject's parents/legal guardian when applicable. They will be provided sufficient time to review the permission/assent/consent form, have all questions answered, and concerns addressed. If they agree to participate, they will sign the permission/assent/consent form.

-Following permission/assent/consent, screening labs will be drawn. If the patient is unable to complete the study labs at this time, a time will be arranged to have these performed at least 1 day prior to Study Drug Day #1. The laboratory evaluation will consist of the following.

1. Research chemistry panel (Sodium, Potassium, Chloride, Carbon Dioxide, Anion Gap, Calcium, Phosphorus, Magnesium, Glucose, BUN, Creatinine, Total Protein, Albumin, Bilirubin, ALT, AST, Alkaline Phosphatase, GGT, LDH, Cholesterol, Uric Acid and Triglyceride) (3 mL blood in mint green or red top with yellow ring gel tube)
2. Complete blood count with differential (1 mL in a 3 mL EDTA lavender top tube or 250 uL in a microtainer)
3. Creatine phosphokinase (0.2ml in gel mint green or red top w/ gold ring)
4. C-reactive protein (1 ml of blood in a mint green or red top tube w/ yellow ring gel; or EDTA).

   -If the patient is currently taking a statin, they will be asked to discontinue this agent until after the completion of the entire study.

   -Finally, scheduling of the subsequent study days will take place at this visit. Study Drug Day #1 will be scheduled 6 days and up to 14 days following the screening visit. Study Drug Day #2 will be scheduled 6 days and up to 14 days following Study Drug Day #1.

   Drug Study Day #1 (Approximately 10 hours) -Upon arrival to the Children's Mercy Hospital Clinical Research Unit, the subject will have a screening physical examination including Tanner staging. For females, a urine specimen will be obtained for beta-human chorionic gonadotropin pregnancy test.

   -Once cleared to participate, the subject will have an indwelling, silastic cannula (21 or 24 Ga) placed in a peripheral vein on the hand or forearm for the purpose of repeated blood sampling to support the pharmacokinetic aims of the study. Patency of this cannula will be maintained throughout the study period using a sterile solution of heparinized saline.

   -A single oral dose of either simvastatin or pravastatin will be ingested with 150ml of tap water after an overnight fast. The sequence of statin administered will be randomized between the two study visits. For two hours following study article administration, subjects will remain fasted with only small sips of water permitted. A standard, age-appropriate heart healthy meal will be served 2 hours after statin administration and a snack will be served in the afternoon of the study day. Water will be permitted ad libitum.
   * In the event that the patient vomits within 2 hours of ingestion of Study Drug Day #1, they will be withdrawn from the study for that day and rescheduled. The subject will be rescheduled up to 14 days after the screening visit. If they are unable to be rescheduled within 14 days of the original screening labs, the labs will be redrawn that day. In the event that the patient vomits within 2 hours of ingestion of Study Drug Day #2, they will be withdrawn from the study for that day and rescheduled. The subject can be rescheduled 6 days and up until 14 days after Study Drug Day #1. If a more than 14 days, but no more than 21 days have transpired since Study Drug Day#1, the subject can be rescheduled, but must have repeated screening labs performed.
   * Serial venous blood samples (1.5 ml each) will be drawn from the indwelling venous cannula to measure plasma drug and drug metabolite levels of the ingested drug before ingestion (time 0), and at 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours post ingestion. Should the patency of the indwelling cannula be lost, it will either be placed or alternatively, remaining blood samples will be obtained by sterile venipuncture at the desire of the study subject. After the samples are drawn, they will be placed into glass tubes containing potassium EDTA and gently mixed by repeated inversion. They will then be immediately centrifuged at 4ºC for a total of 10 minutes at 600g (~2000RPM) and will immediately be placed in an ice bath to be transported to the Clinical Pharmacology Laboratory where they will be processed. The cellular component of the time 0 samples will be retained for future isolation of leukocyte DNA. The plasma component of each of the repeated blood sample obtained to support the pharmacokinetic objectives of the study will be removed by manual aspiration and transferred to a labeled, polypropylene cryovial which will be placed at -80ºC where it will be stored until analysis.
   * Once the 8 hour post-dose sample is taken, blood (5.2 ml) for study safety labs will be drawn, the IV cannula will be removed, and the patient will be discharged from the Clinical Pharmacology unit after the Drug Study Day #2 is confirmed with the study subject and/or subject's parent(s).

   Drug Study Day #2 (Approximately 10 hours) -Following a minimum of 6 days and up to 14 days after the first drug ingestion day (wash out period), the subject will brought back to the CMH Clinical Research Unit for another single dose pharmacokinetic study. Following a physical examination and insertion of a peripheral IV cannula, the alternate statin that was not administered on the first drug study day will be given with 150 ml tap water after an overnight fast. The same blood sampling scheme will be used as described for study day #1. Blood for study safety labs will be obtained after the last drug level sample is drawn and the patient will then be discharged from the CMH Clinical Research Unit. The total amount of blood required for the entire study is summarized in the following table.

   Study Day Amount of Blood Screening Visit 5.2ml (Screening Labs) Drug Study Day #1 13.5ml (PK study labs) 5.2ml (Safety labs) Drug Study Day #2 13.5ml (PK study labs) 5.2ml (Safety labs)

   Total 42.6ml (Over a 1 month period of time)

   One week after completion of Drug Study Day #2 or in the event of early withdrawal, the family will be contacted via telephone to screen for post-study adverse events as defined section 5.

   1.10. Randomization The proposed study is a single-dose pharmacokinetic study comparing two statin drugs, simvastatin and pravastatin. The sequence of administration of the two statins will be randomized for each study participant.

   The Children's Mercy Hospital Investigational Drug Service (IDS) Pharmacy will be responsible for the randomization procedure and will maintain control of the sequence randomization. This is an open label study, so neither the investigators nor subjects will be blinded to the sequence randomization.

2. Laboratory Evaluation 2.1. Drug and Metabolite Analysis After ingestion of a single statin dose, the corresponding drug and its metabolites will be quantified. Pravastatin is administered in its active, open acid form and does not have any significantly active metabolites 27. The most common inactive metabolite isolated in plasma is 3'α-isopravastatin and it is formed non-enzymatically primary in the acidic conditions of the stomach 53. Therefore, after pravastatin ingestion, serial plasma levels of pravastatin acid and 3'alpha-isopravastatin will be assessed. (Additional details of plasma sampling intervals are outlined in Section 1.9). Simvastatin is administered in its inactive, lactone form and undergoes hydrolysis to the major active metabolite which is beta-hydroxy simvastatin acid. Minor metabolites are 6'-hydroxy-simvastatin, 3'hydroxy-simvastatin, 3''-hydroxy-simvastatin, 6'exomethylene-simvastatin, 6'-hydroxymethyl-simvastatin, and 6'-hydroxycarbonyl-simvastatin 25. Several of these metabolites, when converted to their acid forms, have reported activities in dogs but seem to accumulate in the bile with little detectable in plasma 54. Therefore, in this study, only serial plasma levels of simvastatin and simvastatin acid will be assessed. (Additional details of plasma sampling intervals are outlined in Section 5.0).

Analytical strategies for the determination of simvastatin and simvastatin acid:

Simvastatin and simvastatin acid will be determined using a high-throughput salting-out assisted liquid/liquid extraction (SALLE) method with acetonitrile and mass spectrometry compatible salts for simultaneous LC-MS/MS analysis as previously described 55. This method has been extensively validated according to FDA guidelines, and more importantly, demonstrates minimal interconversion of simvastatin and simvastatin acid during sample preparation. A brief outline of the method is as follows. Plasma samples will be thawed at 4ºC in a temperature-controlled water bath, and kept at this temperature during the procedure to minimize analyte interconversion. To an aliquot of sample, a stable deuterated isotope-labeled internal standard of simvastatin and simvastatin acid (Toronto Research Chemicals) are added to allow stable isotope dilution mass spectrometry. The sample is then extracted by the SALLE procedure at pH 4.5 to minimize the interconversion of simvastatin between the lactone and acid form. The extract is stable in the autosampler for 33 hours at 4ºC, and will be analyzed by LC-MS/MS within this timeframe. Sample analysis will occur on a Waters TQ-S triple quadupole mass spectrometer coupled to a Waters Acquity Ultra Performance Liquid Chromatograph (UPLC-MS-MS), utilizing the chromatographic conditions (including column) as previously described 55. Simvastatin and its internal standard will be monitored in positive ion-mode utilizing the 450-285 and 453-285 transitions of the methyl ammonium adducts respectively. Simvastatin acid and its internal standard will be measured in negative ion-mode due to poor ionization in positive mode. Transitions for these analytes will be 435-319 and 438-319. All plasma samples will be run in duplicate for each sampling time interval to assure validity. The remaining plasma not used in the analysis will be stored within the Clinical Pharmacology laboratory in dedicated freezers/refrigerators as outlined in the CPR Repository. Use of these samples for further study will be at the discretion of the CPR director as outlined in the CPR protocol (CMH IRB# 12040220).

Analytical strategies for the determination of pravastatin and pravastatin lactone:

A large number of analytical strategies for the determination of pravastatin and pravastatin lactone have been described in the literature 56-59, however many of these are labor intensive and not as high throughput as the methodology presented for simvastatin. Due to the structural similarities between simvastatin and pravastatin it is highly likely that the analytical method for simvastatin can be adapted for the analysis of pravastatin and pravastatin lactone with minimal change. In the unlikely event that the simvastatin method cannot be adapted to pravastatin and pravastatin lactone analysis, we will utilize the method presented by Vlckova et al 60.

3 Assessment of Pharmacokinetics 3.1 Pharmacokinetic Parameters Pharmacokinetic analyses will be conducted using Kinetica version 5.0 (Thermo Electron, Philadelphia, PA). Pravastatin, simvastatin, and metabolite plasma concentration vs. time data will be curve fit using a peeling algorithm to generate initial monoexponential parameter estimates. Final estimates of the terminal elimination rate constant (delta z) will be determined from an iterative, linear least squares regression algorithm. A model-independent approach will be used and parameters of interest determined as follows. Individual Cmax and Tmax will be obtained by direct examination of the plasma concentration versus time profile. The area under the plasma concentration versus time curve during the sampling period (AUC0-n) will be calculated using the mixed log-linear method where n refers to the final sampling time with quantifiable drug or metabolite concentrations. Extrapolation of the AUC to infinity (AUC0-infinity) will be achieved by the summation of AUC0-n + Cpn/delta z, where Cpn is the last observable plasma concentration calculated from the curve fit of the terminal slope of the plasma concentration vs. time curve and delta z is the apparent terminal elimination rate constant. Absorption and elimination half-life (t½) will be calculated from the initial and terminal portions of the plasma concentration vs. time curve for each analyte of interest. In the case of metabolites, the corresponding half life term will be that used to denote metabolite formation.

4 Statistical Plan 4.1 Statistical Methods Pravastatin and simvastatin pharmacokinetic data for the study cohort will be examined initially using standard descriptive statistics (i.e., arithmetic mean, geometric mean, standard deviation, coefficient of variation, 95% confidence limits). A repeated measures analysis of variance model will be employed to determine treatment, period, and sequence effects for the resultant primary and secondary pharmacokinetic parameter estimates. Pharmacokinetic parameters reflective of exposure (Cmax, AUC0-n, AUC0-infinity) will be log-transformed using the natural logarithm, the 90% confidence intervals for the difference in the means calculated and the antilog of the confidence limits evaluated against the pre-established bioequivalence criteria as defined in our power calculations. The significance limit accepted for all statistical analyses will be alpha = 0.05.

The contribution of different alleles to variation in the pharmacokinetic parameters of pravastatin and simvastatin will be investigated with multiple regression analysis. The genotype class (non-carriers and carriers) will be treated as independent variables. For Aim #1, the pharmacokinetic variables for each drug will be compared between non-carriers and carriers of variant alleles using independent t-test. Similarly, for Aim #2, the ratio of each pharmacokinetic parameter in carriers to non-carriers (e.g. AUCcarrier/AUCnon-carrier) for pravastatin will be compared to the corresponding ratios following simvastatin administration. All analyses will be performed in SPSS version 18.0 (SPSS, Chicago, IL).

4.2 Subject Population(s) for Analysis Previously studies have shown that highly hydrophilic statins, such as pravastatin, are more dependent on the OATP1B1 transporter compared to more lipophilic statins, such as simvastatin 41, 45. It is theorized that the upstream promoter region (-11187) might have a more pronounced impact on the genotype-phenotype relationship as seen in the previous pediatric study 49. Therefore, our study will be powered to observe a dose-exposure difference in -11187 allelic variants and wild-type/wild-type with pravastatin.

There are anticipated to be 150 subjects enrolled in the CPR database meeting inclusion criteria. The frequency of SLCO1B1 SNPs (-11187G>A, 7-8%) from previous adult studies 61, suggests approximately ~19-22 heterozygous subjects (according to the Hardy Weinberg Equation) in the anticipated number of participants from the CPR database. With a 90% participation/10% attrition rate, there would be ~17-20 subjects.

On the basis of previous data on the adult pharmacokinetics of pravastatin in the variant alleles described above 45, a sample size of 18 in each group (-11187G>A genotype and wild-type control) will have 80% power to detect a difference in means of -101.0 in AUC (0-∞) (the difference between a Group 1 mean, m1, of 102.7 and a Group 2 mean, m2, of 203.7, which is nearly a 2-fold difference) assuming that the Group 1 standard deviation, s1, is 69.1 and the Group 2 standard deviation, s2, is 126.4 using a two group Satterthwaite t-test with a 0.050 two-sided significance level.

Therefore, our target sample size is 18 subjects with SLCO1B1 -11187G>A allele. With age- and sex-matched controls, the total sample size is 36 subjects.

5. Adverse Events An adverse event is defined as any unintended change in the body structure (signs) or body function (symptoms), whether or not considered drug-related. During the entire duration of the study, subjects will be instructed to report all adverse events. All adverse events, whether volunteered, elicited, or noted on physical examination, will be recorded throughout the study, (i.e., from the time of the first dose administration on Day 1 up to 1 week after the entire study completion or subject withdrawal from the study). The severity of adverse events will be categorized as mild, moderate, or severe according to FDA guidelines.

The Investigator will make a determination of the relationship of the adverse event to the study drug using a four-category system (not related, unlikely, suspected, and probable) according to FDA guidelines. A serious adverse drug experience is any adverse test material event occurring at any dose that results in any of the outcomes defined by the FDA.

An unexpected adverse experience is any adverse experience that is not identified in nature, severity, or frequency in the current approved drug labeling or elsewhere in the general investigational plan. Any serious and unexpected adverse clinical event, whether or not related to the study drug, will be reported verbally to the primary investigators within 24 hours of notification.

Subsequently, a Serious Adverse Event (SAE) Report Form will be completed and Children's Mercy Hospital and Clinics Institutional Review Board (IRB) will be notified. A statement from the Principal Investigator outlining the details of the adverse reaction will accompany this form. Laboratory reports and other safety reports will be forwarded as they become available.

NOTE: The term "severe" is often used to describe the intensity (severity) of a specific event (as in mild, moderate, or severe myocardial infarction); the event itself, however, may be of relatively minor medical significance (such as a severe headache). This is not the same as "serious," which is based on participant/event outcome or action criteria usually associated with events that pose a threat to the participant's life or functioning. Seriousness (not intensity) serves as a guide for defining regulatory reporting obligations.

Ethical aspects This study will be conducted according to US and international standards of Good Clinical Practice (FDA regulations 21 CFR 312 for IND studies and FDA guidance E6) for all studies. Applicable government regulations and University of Missouri-Kansas City/Children's Mercy Hospital and Clinics research policies and procedures will also be followed.

This protocol and any amendments will be submitted to the Children's Mercy Hospital and Clinics Institutional Review Board (IRB) for formal approval to conduct the study. The decision of the IRB concerning the conduct of the study will be made in writing to the investigator.

All subjects and parent/legal guardians, when applicable, will be provided a permission/assent/consent form describing this study and providing sufficient information for subjects to make an informed decision about their participation in this study. This consent form will be submitted with the protocol for review and approval by the IRB. Formal consent/permission/assent will be obtained, using the IRB-approved forms, before a subject is submitted to any study procedure. The consent/permission/assent form must be signed by the subject or legally acceptable surrogate, and the investigator-designated research professional obtaining the consent.

ELIGIBILITY:
Inclusion Criteria:

1. Children 8-21 years of age
2. LDL cholesterol >130mg/dl (>95% percentile)
3. Successfully genotyped for SLCO1B1
4. Willing to sign the assent/permission/consent form

Exclusion Criteria:

1. Underlying structural heart disease including congenital heart disease or acquired heart disease.
2. History or laboratory evidence of an underlying intestinal, metabolic, autoimmune, or renal disease that could alter the disposition of simvastatin or pravastatin.
3. Underlying pathology of the gastrointestinal tract or recent surgery which would be expected to alter the rate and/or extent of drug absorption
4. Evidence of previous hypersensitivity to statin medications
5. Unwillingness or inability to have screening labs drawn
6. Refusal to participate in the study
7. Unwillingness or inability to participate in an overnight fast
8. Subjects taking drugs with interactions with statins (CYP3A4 inducers/inhibitors, OATP1B1 inducers/inhibitors)
9. Inability to swallow a tablet drug
10. For females, a positive urine beta-human chorionic gonadotropin pregnancy test result
11. Evidence of hepatic abnormality as determined by values > 3 times the age-specific upper limit of normal for AST, ALT, total and conjugated bilirubin, serum albumin, Alkaline Phosphatase, and GGT.
12. Abnormal red blood cell morphology and/or a hemoglobin less than 9 gm/dl

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2014-06-17 (Actual); Primary Completion 2016-07-05 (Actual); Study Completion 2016-07-05 (Actual)

PRIMARY OUTCOMES:
Evaluate effect of genotype (SLCO1B1) on Cmax pravastatin | 2 years
Evaluate effect of genotype (SLCO1B1) on AUC pravastatin | 2 years
Evaluate effect of genotype (SLCO1B1) on Cmax Simvastatin | 2 years
Evaluate effect of genotype on AUC Simvastatin | 2 years

SECONDARY OUTCOMES:
Evalaute the effect of age on Cmax of pravastatin | 2 years
Evalaute the effect of gender on Cmax of pravastatin | 2 years
Evalaute the effect of race Cmax of pravastatin | 2 years
Evaluate the effect of sexual maturity on Cmax of pravastatin based | 2 years
Evaluate the effect of age on Cmax of simvastatin | 2 years
Evaluate the effect of gender on Cmax of simvastatin | 2 years
Evaluate the effect of race on Cmax of simvastatin | 2 years
Evaluate the effect of sexual maturity on Cmax of simvastatin | 2 years
Evaluate the effect of age on AUC of pravastatin | 2 years
Evaluate the effect of gender on AUC of pravastatin | 2 years
Evaluate the effect of race on AUC of pravastatin | 2 years
Evaluate the effect of sexual maturity on AUC of pravastatin | 2 years
Evaluate the effect of age on AUC of simvastatin | 2 years
Evaluate the effect of gender on AUC of simvastatin | 2 years
Evaluate the effect of race on AUC of simvastatin | 2 years
Evaluate the effect of sexual maturity on AUC of simvastatin | 2 years
Evaluate the effect of age on Ka of pravastatin | 2 years
Evaluate the effect of gender on Ka of pravastatin | 2 years
Evaluate the effect of race on Ka of pravastatin | 2 years
Evaluate the effect of sexual maturity on Ka of pravastatin | 2 years
Evaluate the effect of age on Ka of simvastatin | 2 years
Evaluate the effect of gender on Ka of simvastatin | 2 years
Evaluate the effect of race on Ka of simvastatin | 2 years
Evaluate the effect of sexual maturity on Ka of simvastatin | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

REFERENCES:
- [Derived] Wagner JB, Abdel-Rahman S, Van Haandel L, Gaedigk A, Gaedigk R, Raghuveer G, Kauffman R, Leeder JS. Impact of SLCO1B1 Genotype on Pediatric Simvastatin Acid Pharmacokinetics. J Clin Pharmacol. 2018 Jun;58(6):823-833. doi: 10.1002/jcph.1080. Epub 2018 Feb 22. PMID 29469964